CLINICAL TRIAL: NCT06944782
Title: BREATH: Breakthrough Research in Electromyography for the Assessment of Sleep-disordered BreaTHing
Brief Title: Diagnosing Obstructive Sleep Apnea Using Electromyography of the Muscles of the Mouth
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Powell Mansfield Inc. (Other)
Responsible Party: Principal Investigator, Jejo Koola, Associate Professor of Medicine, University of California, San Diego
Other Study IDs: 315616-00001; R42HL176325-01 (NIH)
Record Dates: First submitted 2025-04-14; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea (OSA); OSA; Healthy Volunteers; Electromyography
Keywords: sleep study; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Adults who have completed a sleep study but were not diagnosed with sleep apnea.
  Interventions: Diagnostic Test: Electromyography (EMG) of the Oropharynx
- People with Sleep Apnea: Adults who have completed a sleep study and were diagnosed with sleep apnea.
  Interventions: Diagnostic Test: Electromyography (EMG) of the Oropharynx

INTERVENTIONS:
Diagnostic Test: Electromyography (EMG) of the Oropharynx — The transmembranous electromyography (tmEMG) probe is a disposable single-use bipolar recording device with the sensor configured with two electrodes located at the distal end of the probe in a parallel orientation. Unlike conventional EMG probes that are designed to be inserted into the muscle, the tmEMG probe is placed on the surface of the muscle similar to a surface electrode; the tip of the probe is approximately the size of a ball point pen, which allows us to record from the smaller muscles inside the mouth. Recordings will be taken from the genioglossus and palatoglossus in the mouth bilaterally. Recordings will be taken while the subject performs various maneuvers such as shallow breathing, deep breathing, and pressing their tongue against the side of their mouth.
  Other Names: transmembranous EMG; tmEMG

SUMMARY:
The investigators will establish how well a novel, quick, and painless way of measuring muscle activity from the mouth and throat works for detecting sleep apnea. This technology is called transmembraneous electromyography (tmEMG). Leveraging two technologies, a new probe capable of recording muscle activity by lightly touching the muscle, as well as a machine learning model for signal interpretation, the investigators will conduct an initial observational feasibility study in phase 1, followed by a larger observational cohort study in phase 2 to assess the performance of deep learning enhanced tmEMG. The study will address a critical unmet need in sleep apnea diagnostics: the availability of an inexpensive, accurate diagnostic test for screening at point of care.

DETAILED DESCRIPTION:
Given night-to-night variability and/or changes in OSA severity over time, study participants will undergo a 2-night home sleep test to verify the results of a prior sleep test as part of our screening activities. After verifying that the results of the home sleep test are concordant with the participant's previously administered clinical sleep study, they will be brought to the study clinic. Participants from both arms will undergo testing of four oropharyngeal muscles: left and right palatoglossus, left and right genioglossus. Using the transmembranous electromyography (tmEMG) probe, recordings will be obtained from each muscle using various provocative maneuvers. For the palatoglossus, recordings will be obtained during normal shallow inspiration as well as deep forceful inspiration. For the genioglossus, recordings will be obtained during maximal voluntary contraction as well sub-maximal voluntary contraction of the tongue against resistance (either the buccal mucosa or the front incisors).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Subject must have completed a prior sleep test.

   1. Subjects may be recruited if the last prior sleep test either determined that they do not have sleep apnea OR they have moderate to severe sleep apnea. No sleep apnea is defined by AHI < 5; moderate to severe sleep apnea is defined by AHI >= 15.
   2. To be fully eligible, the prior test result needs to be verified via 2-night home sleep test (using the average AHI from the 2 nights). If OSA status (i.e., AHI<5/h or >=15/h) from the 2-night HST vs last prior sleep test is discordant, then participants will be excluded as screen failures.

Exclusion Criteria:

1. Current use of OSA therapy, including PAP (positive airway pressure) or non-invasive ventilation on a daily basis
2. Prior uvulopalatopharyngoplasty surgery for sleep apnea.
3. Inability to install WatchPAT ONE application on smartphone or tablet or unwillingness/inability to use the WatchPAT ONE home sleep study device
4. Prisoners are excluded due to ethical, legal, and practical concerns
5. Individuals who are pregnant are excluded due to temporary changes in habitus, fluid shifts, and potential changes to oropharyngeal musculature may impact tmEMG assessment. This important subpopulation will be investigated in a later phase study.
6. Inability to stop tobacco, marijuana, or vaping on the day of testing.
7. Binge alcohol use behaviors (4+ drinks on the same occasion on 5+ days in the past month).
8. Medication use that may cause central apnea that in the judgment of the investigators could impact the safety or results of the study
9. Allergy to benzocaine topical anesthetic or other ester class local anesthetics (lidocaine, etc.)
10. Current psychiatric illness other than treated mood disorders
11. Unable or unwilling to provide informed consent or comply with research procedures
12. Active Cancer due to potential interference with study results
13. Major comorbidities which in the judgment of the investigators could impact the safety or results of the study
14. Inability to sign consent and participate in the study in English. This study involves use of an investigational device; the technical nature of the study and the consenting process and consent form make it impractical to include subjects who cannot participate in English.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited from adult patients who have undergone a sleep study, generally within San Diego County.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
AUC (Area Under the Curve) | 3 months
  Diagnostic accuracy, as measured by the area under the receiver operator characteristic curve (AUC), of DL-tmEMG algorithm in detecting moderate to severe OSA.

SECONDARY OUTCOMES:
Delta AUC When Adding Clinical Data | 3 months
  The secondary outcome is to assess the incremental improvement in diagnostic performance, as measured by the change in AUC, when selected clinical variables are incorporated into the tmEMG-based machine learning model. These clinical variables may include demographic characteristics, sleep-related questionnaire scores (e.g., STOP-Bang, Epworth Sleepiness Scale), and relevant medical history. Model performance with and without clinical variables will be compared using appropriate statistical techniques to evaluate the added predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Jejo Koola, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No